CLINICAL TRIAL: NCT04736355
Title: DAOIB for the Treatment of Mild Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201800387A3
Record Dates: First submitted 2021-01-31; First posted 2021-02-03 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAOIB (Experimental): oral, for 24 weeks
  Interventions: Drug: DAOIB
- Placebo (Placebo Comparator): oral, for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DAOIB — oral, for 24 weeks
  Arms: DAOIB
Drug: Placebo — oral, for 24 weeks
  Arms: Placebo

SUMMARY:
NMDA neurotransmission plays an important role in learning and memory. NMDA receptor-enhancing agent improved the cognitive function of patients with early-phase Alzheimer's disease. This study is a randomized, double-blind, placebo-controlled drug trial. All subjects will be allocated randomly to 2 groups: (1) DAOIB group; (2) placebo group. The study period is 24 weeks. The investigators hypothesize that DAOIB may yield better efficacy than placebo for cognitive function in patients with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild cognitive impairment
* MMSE between 17-26
* CDR 0.5

Exclusion Criteria:

* Hachinski Ischemic Score > 4
* Substance abuse/dependence
* Parkinson disease, epilepsy, dementia with psychotic features
* Major psychiatric disorders
* Major physical illnesses
* Severe visual or hearing impairment

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's disease assessment scale - cognitive subscale at week 8, 16 and 24 | week 0, 8, 16, 24
  Alzheimer's disease assessment scale-cognitive subscale consists of 11 tasks. Its scores range from 0 (best) to 70 (worst).

SECONDARY OUTCOMES:
Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24 | week 8, 16, 24
  Clinician's Interview-Based Impression of Change plus Caregiver Input score is a global assessment of change based on a comprehensive, semi-structured interview which includes caregiver-supplied information. It is a 7-point rating scale ranging from 1-7, where 1 represents markedly improved; 4, no change; and 7, markedly worse.
Change from baseline in Alzheimer's disease Cooperative Study scale for ADL in MCI (ADCS-MCI-ADL) score at week 8, 16 and 24 | week 0, 8, 16, 24
  ADCS-MCI-ADL appears to be a suitable instrument for evaluating activities of daily living in mild cognitive impairment. Its scores range from 0 (worst) to 78 (best).
Change from baseline in Medical Outcomes Study Short-Form-36 (SF-36) score at week 8, 16 and 24 | week 0, 8, 16, 24
  The SF-36 consists of eight sections which assess the quality of life.
Change from baseline in the composite score of a battery of additional cognitive tests at week 8, 16 and 24 | week 0, 24
  The battery of additional cognitive tests include speed of processing (Category Fluency), working memory (verbal and nonverbal, Wechsler Memory Scale), learning and memory tests (verbal and visual, Wechsler Memory Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin CH, Wang SH, Lane HY. Sodium benzoate, a D-amino acid oxidase inhibitor, improved short-term memory in patients with mild cognitive impairment in a randomized, double-blind, placebo-controlled clinical trial. Psychiatry Clin Neurosci. 2025 Aug;79(8):466-472. doi: 10.1111/pcn.13841. Epub 2025 May 23. PMID 40405827